CLINICAL TRIAL: NCT04572243
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study With Open-Label Extension Phase of Lorcaserin as Adjunctive Treatment in Subjects With Dravet Syndrome
Brief Title: A Study of Lorcaserin as Adjunctive Treatment in Participants With Dravet Syndrome
Acronym: MOMENTUM 1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated by Sponsor and the decision was not due to any safety or efficacy reasons.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2023-A001-304
Expanded Access: NCT04457687 (Available)
Record Dates: First submitted 2020-09-30; First posted 2020-10-01 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-01

CONDITIONS: Epilepsies, Myoclonic
Keywords: Dravet Syndrome; Lorcaserin; E2023; Epilepsy; Seizures
MeSH Terms: conditions — Epilepsies, Myoclonic; Epilepsy; Seizures | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lorcaserin (Core Study and Open-label Extension Phase) (Experimental): Participants will be randomized to receive lorcaserin administered as an oral suspension, twice daily for 14 weeks during the core treatment period. Dose will be based on body weight as follows: target dose for participants weighing 10 to less than (<) 20, 20 to <40, and greater than or equal to (>=) 40 kilogram (kg) will be 5, 10, and 20 milligram per day (mg/day) respectively. Based on clinical response and tolerability and within 2 weeks of treatment, dose can be increased up to 10, 20 mg/day for participants weighing 10 to <20, 20 to <40 kg respectively. Participants completing the core treatment period will enter a 12-week extension phase and will receive lorcaserin.
  Interventions: Drug: Lorcaserin
- Placebo (Core Study) + Lorcaserin (Open-label Extension Phase) (Placebo Comparator): Participants will be randomized to receive lorcaserin matching placebo administered as an oral suspension, twice daily for 14 weeks during the core treatment period. Dose will be based on body weight as follows: target dose for participants weighing 10 to <20, 20 to <40, and >=40 kg will be 5, 10, and 20 mg/day respectively. Based on clinical response and tolerability and within 2 weeks of treatment, dose can be increased up to 10, 20 mg/day for participants weighing 10 to <20, 20 to <40 kg respectively. Participants completing the core treatment period will enter a 12-week extension phase and will receive lorcaserin.
  Interventions: Drug: Placebo; Drug: Lorcaserin

INTERVENTIONS:
Drug: Placebo — Placebo matching to lorcaserin oral tablet, administered as oral suspension.
  Arms: Placebo (Core Study) + Lorcaserin (Open-label Extension Phase)
Drug: Lorcaserin — Lorcaserin oral tablet, administered as oral suspension.
  Other Names: E2023

SUMMARY:
The primary purpose of the study is to demonstrate that lorcaserin has superior efficacy compared to placebo on percent change in frequency of convulsive seizures per 28 days in participants with Dravet syndrome.

ELIGIBILITY:
Key Inclusion Criteria:

Participants must meet all of the following criteria to be included in this study:

1. Male or female, age 2 years and older at the time of informed consent
2. Diagnosis of epilepsy with Dravet syndrome
3. Has at least 4 convulsive seizures during the 4 weeks of baseline
4. Current treatment with antiepileptic drugs must be stable for at least 4 weeks before screening, and be expected to remain stable throughout the study

Key Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this study:

1. Use of lorcaserin within 4 weeks before screening, or any history of it being discontinued due to lack of efficacy or adverse reactions
2. Use of fenfluramine within 2 months before screening, any history of lack of fenfluramine efficacy, or any history of valvulopathy at baseline with history of fenfluramine use
3. Recent or concomitant use of serotonergic medications or monoamine oxidase inhibitors
4. Presence of progressive central nervous system disease other than Dravet syndrome

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (25):
  - Children's of Alabama / University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Los Angeles (UCLA), Los Angeles, California
  - UCSD Rady's Children's Hosptial, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Northwest Florida Clinical Research Group, Gulf Breeze, Florida
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Miami Children's Hospital - Nicklaus Children's Hospital, Miami, Florida
  - Pediatric Neurology, P.A., Winter Park, Florida
  - Rare Disease Research Center Pediatrics, LLC, Atlanta, Georgia
  - Mid-Atlantic Epilepsy and Sleep Center - Bethesda, Bethesda, Maryland
  - Spectrum Health/ Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - University of Missouri, Department of Child Health, Division of Neurology, Columbia, Missouri
  - Institute of Neurology and Neurosurgery at Saint Barnabas, Livingston, New Jersey
  - Northwell Health - Neuroscience Institute at Great Neck, New Hyde Park, New York
  - NYU Langone Comprehensive Epilepsy Center, New York, New York
  - New York Medical College, New York, New York
  - NorthWell Health - Lennox Hill Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Hospital Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Children's Hospital - VH, London Health Sciences Centre, London, Ontario
  - University of Toronto Division of Hematology Oncology/The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 15 investigative sites in Canada and the United States from 23 September 2020 to 15 August 2024.
Pre-assignment Details: The study was conducted in two phases (Core Study and an Open-label Extension Phase). A total of 27 participants were screened, of which 5 were screen failures and 22 were enrolled to receive study treatment. This study was terminated due to sponsor decision, and not due to safety concerns. As pre-planned, the data collection and analysis were based on treatments (placebo or lorcaserin) in Core Study and Extension Phase. The dose level wise data was not collected in this study.
Groups:
- Core Study: Placebo: Participants received lorcaserin-matching placebo, oral suspension, twice daily for 14 weeks.
- Core Study: Lorcaserin: Participants weighing 10 to less than (<) 20 kilogram (kg), 20 to <40 kg, and greater than or equal to (>=) 40 kg received lorcaserin oral suspension, at dose of 5 milligrams per day (mg/day), 10 mg/day, and 20 mg/day, respectively. During the first 2 weeks of the treatment, depending on the participant's clinical response and tolerability, the dose was increased up to 10 mg/day for participants weighing 10 to <20 kg and up to 20 mg/day for those weighing 20 to <40 kg and >=40 kg. The total treatment duration in Core Study was 14 weeks.
- Extension Phase: Placebo Then Lorcaserin: Participants who received placebo in Core Study and entered Extension Phase, received lorcaserin, oral suspension based on body weight as the target dose for participants weighing 10 to <20 kg, 20 to <40 kg, and >=40 kg was 5 mg/day, 10 mg/day, and 20 mg/day, respectively for first 6 weeks in Extension Phase. Based on clinical response and tolerability, the dose was increased up to 10 mg/day for participants weighing 10 to <20 kg and up to 20 mg/day for those weighing 20 to <40 kg and >=40 kg for second 6 weeks in Extension Phase. The total treatment duration in Extension Phase was 12 weeks.
- Extension Phase: Lorcaserin: Participants who received lorcaserin in Core Study and entered Extension Phase, received lorcaserin at the same dose they were receiving at end of Core Study for first 6 weeks in Extension Phase. Based on clinical response and tolerability, the dose increased up to 10 mg/day for participants weighing 10 to <20 kg and up to 20 mg/day for those weighing 20 to <40 kg and >=40 kg during second 6 weeks in Extension Phase. The total treatment duration in Extension Phase was 12 weeks.
Period: Core Study: 14 Weeks
Arm/Group | Core Study: Placebo | Core Study: Lorcaserin | Extension Phase: Placebo Then Lorcaserin | Extension Phase: Lorcaserin
Started | 11 | 11 | 0 | 0
Treated | 10 | 11 | 0 | 0
Completed | 8 | 7 | 0 | 0
Not Completed | 3 | 4 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Subject choice | 0 | 2 | 0 | 0
Not completed — Withdrawal of consent | 1 | 0 | 0 | 0
Not completed — Randomized but not treated | 1 | 0 | 0 | 0
Period: Extension Phase: 12 Weeks
Arm/Group | Core Study: Placebo | Core Study: Lorcaserin | Extension Phase: Placebo Then Lorcaserin | Extension Phase: Lorcaserin
Started | 0 | 0 | 7 (Participants who completed the Core Study, received treatment in Extension Phase. However, one participant who received placebo and completed the Core Study did not continue in Extension Phase due to unspecified reason.) | 7
Completed | 0 | 0 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Groups:
- Placebo/ Lorcaserin: Participants received lorcaserin-matching placebo, oral suspension, twice daily for 14 weeks in Core Study followed by lorcaserin, oral suspension based on body weight as the target dose for participants weighing 10 to <20 kg, 20 to <40 kg, and >=40 kg was 5 mg/day, 10 mg/day, and 20 mg/day, respectively for first 6 weeks in Extension Phase. Based on clinical response and tolerability, the dose was increased up to 10 mg/day for participants weighing 10 to <20 kg and up to 20 mg/day for those weighing 20 to <40 kg and >=40 kg for second 6 weeks in Extension Phase. The total treatment duration in Core Study was 14 weeks and 12 weeks in Extension Phase.
- Lorcaserin/ Lorcaserin: Participants weighing 10 to <20 kg, 20 to <40 kg, and >=40 kg received lorcaserin oral suspension, at dose of 5 mg/day, 10 mg/day, and 20 mg/day, respectively in Core Study. During the first 2 weeks of the treatment, depending on the participant's clinical response and tolerability, the dose was increased up to 10 mg/day for participants weighing 10 to <20 kg and up to 20 mg/day for those weighing 20 to <40 kg and >=40 kg. During Extension Phase, participants continued the same dose of Core Study for first 6 weeks in Extension Phase. Based on clinical response and tolerability, the dose increased up to 10 mg/day for participants weighing 10 to <20 kg and up to 20 mg/day for those weighing 20 to <40 kg and >=40 kg during second 6 weeks in Extension Phase. The total treatment duration in Core Study was 14 weeks and 12 weeks in Extension Phase.
- Total: Total of all reporting groups
Arm/Group | Placebo/ Lorcaserin | Lorcaserin/ Lorcaserin | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: year] | 12.9 (10.32) | 12.7 (7.71) | 12.8 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 7 | 10 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Core Study: Percent Change From Baseline in Convulsive Seizure Frequency Per 28 Days During the Treatment Period
Description: Seizure frequency for convulsive seizures was based on number of seizures per 28 days, calculated during the baseline period (Week -4 to Week 0) and 14-week treatment period, as the number of seizures during each respective period divided by the number of non-missing days during each respective period, multiplied by 28. Percent change from baseline was calculated as: ([post-baseline value minus the baseline value] / baseline value) *100.
Time Frame: Baseline up to Week 14
Population: The FAS was the group of randomized participants who received at least 1 dose of study drug and had at least 1 post-dose primary efficacy measurement.
Measure: Median (Full Range); unit: percent change
Groups:
- Core Study: Lorcaserin: Participants weighing 10 to <20 kg, 20 to <40 kg, and >=40 kg received lorcaserin oral suspension, at dose of 5 mg/day, 10 mg/day, and 20 mg/day, respectively. During the first 2 weeks of the treatment, depending on the participant's clinical response and tolerability, the dose was increased up to 10 mg/day for participants weighing 10 to <20 kg and up to 20 mg/day for those weighing 20 to <40 kg and >=40 kg. The total treatment duration in Core Study was 14 weeks.
Arm/Group | Core Study: Placebo | Core Study: Lorcaserin
Number analyzed (Participants) | 10 | 10
percent change | 18.78 [-53.7 to 131.5] | -78.88 [-100.0 to 542.9]
Statistical Analysis 1: Comparison: Core Study: Placebo vs Core Study: Lorcaserin; Test type: Superiority; Median Difference (Final Values) = -86.08, 95% CI 2-sided [-144.01 to -28.14]

2. Secondary Outcome: Core Study: Percentage of Participants With 50% or Greater Response for Convulsive Seizures in the Treatment Period Compared to Baseline
Description: A responder was defined as a participant who experienced a reduction of 50% or greater in the frequency of convulsive seizures during the 14-week treatment period compared to the baseline period (Week -4 to Week 0). Seizure frequency was based on number of seizures per 28 days, calculated during the baseline period (Week -4 to Week 0) and treatment period, as the number of seizures during each respective period divided by the number of non-missing days during each respective period, multiplied by 28.
Time Frame: Baseline up to Week 14
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Study: Placebo | Core Study: Lorcaserin
Number analyzed (Participants) | 10 | 10
percentage of participants | 20.0 | 60.0
Statistical Analysis 1: Comparison: Core Study: Placebo vs Core Study: Lorcaserin; Test type: Superiority; Odds Ratio (OR) = 6.0, 95% CI 2-sided [0.81 to 44.35]

3. Secondary Outcome: Core Study: Percentage of Participants Who Were Free From Convulsive Seizures in the Treatment Period
Description: A responder was a participant who experienced a 100% reduction (seizure freedom) in convulsive seizure frequency in the 14-week treatment period relative to the baseline period (Week -4 to Week 0). Seizure frequency was based on number of seizures per 28 days, calculated during the baseline period (Week -4 to Week 0) and treatment period, as the number of seizures during each respective period divided by the number of non-missing days during each respective period, multiplied by 28.
Time Frame: Baseline up to Week 14
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Study: Placebo | Core Study: Lorcaserin
Number analyzed (Participants) | 10 | 10
percentage of participants | 0.0 | 10.0

4. Secondary Outcome: Core Study: Plasma Concentrations of Lorcaserin
Description: Plasma Concentrations of Lorcaserin was evaluated and reported.
Time Frame: Weeks 1, 2, 6, 15: Pre-dose and 1 to 2 hours post-dose; Weeks 4,10: Pre-dose, 1 to 2 hours and 3 to 6 hours post-dose
Population: The Pharmacokinetic (PK) analysis set was the group of all randomized participants from whom at least measurable lorcaserin plasma concentration was obtained with associated documented dosing history. Here 'n' refers to number of participants analyzed at different timepoints for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Core Study: Lorcaserin
Number analyzed (Participants) | 7
nanograms per milliliter (ng/mL)
  Week 1: Pre-dose: number analyzed (Participants) | 1
  Week 1: Pre-dose | 52.0 (NA) — Standard deviation could not be derived as the analysis was based on a single participant
  Week 1: 1 to 2 hours post-dose: number analyzed (Participants) | 1
  Week 1: 1 to 2 hours post-dose | 106 (NA) — Standard deviation could not be derived as the analysis was based on a single participant
  Week 2: Pre-dose: number analyzed (Participants) | 5
  Week 2: Pre-dose | 22.1 (14.5)
  Week 2: 1 to 2 hours post-dose: number analyzed (Participants) | 5
  Week 2: 1 to 2 hours post-dose | 32.7 (22.7)
  Week 4: Pre-dose: number analyzed (Participants) | 2
  Week 4: Pre-dose | 48.5 (13.2)
  Week 4: 1 to 2 hours post-dose: number analyzed (Participants) | 2
  Week 4: 1 to 2 hours post-dose | 107 (76.9)
  Week 4: 3 to 6 hours post-dose | 60.5 (36.0)
  Week 6: Pre-dose: number analyzed (Participants) | 4
  Week 6: Pre-dose | 22.7 (11.8)
  Week 6: 1 to 2 hours post-dose: number analyzed (Participants) | 4
  Week 6: 1 to 2 hours post-dose | 41.0 (20.6)
  Week 10: Pre-dose: number analyzed (Participants) | 1
  Week 10: Pre-dose | 32.9 (NA) — Standard deviation could not be derived as the analysis was based on a single participant
  Week 10: 1 to 2 hours post-dose: number analyzed (Participants) | 1
  Week 10: 1 to 2 hours post-dose | 52.4 (NA) — Standard deviation could not be derived as the analysis was based on a single participant
  Week 10: 3 to 6 hours post-dose | 66.7 (33.7)
  Week 15: Pre-dose: number analyzed (Participants) | 1
  Week 15: Pre-dose | 33.6 (NA) — Standard deviation could not be derived as the analysis was based on a single participant
  Week 15: 1 to 2 hours post-dose: number analyzed (Participants) | 1
  Week 15: 1 to 2 hours post-dose | 31.4 (NA) — Standard deviation could not be derived as the analysis was based on a single participant

5. Secondary Outcome: Core Study: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event (AE) that emerges during treatment, was absent at pretreatment (baseline) or reemerges during treatment, was present at pretreatment (baseline) but stopped before treatment or worsens in severity during treatment relative to the pretreatment state, when the AE was continuous. An AE was any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE did not necessarily have a causal relationship with the medicinal product.
Time Frame: From first dose of study drug up to end of 4 weeks of follow up after last dose of study drug (up to Week 18)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Core Study: Placebo | Core Study: Lorcaserin
Number analyzed (Participants) | 10 | 11
Participants | 7 | 9

ADVERSE EVENTS:
Time Frame: Core Study: From first dose of study drug up to end of 4 weeks of follow up after last dose of study drug (up to Week 18); Extension Phase: From first dose of study drug in Extension Phase (Week 15) up to end of 4 weeks of follow up after last dose of study drug (up to Week 30)
Description: The Safety Analysis Set was the group of participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Arm/Group | Core Study: Placebo | Core Study: Lorcaserin | Extension Phase: Placebo Then Lorcaserin | Extension Phase: Lorcaserin
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/11 | 0/7 | 1/7
Other Adverse Events (participants affected / at risk) | 7/10 | 8/11 | 4/7 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Study: Placebo (N=10) | Core Study: Lorcaserin (N=11) | Extension Phase: Placebo Then Lorcaserin (N=7) | Extension Phase: Lorcaserin (N=7)
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Study: Placebo (N=10) | Core Study: Lorcaserin (N=11) | Extension Phase: Placebo Then Lorcaserin (N=7) | Extension Phase: Lorcaserin (N=7)
Dacryostenosis acquired (Eye disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Body temperature decreased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0
Sluggishness (General disorders) | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated due to sponsor decision, and not due to safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT04572243/Prot_002.pdf
  • Statistical Analysis Plan (2024-05-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT04572243/SAP_003.pdf